CLINICAL TRIAL: NCT01431040
Title: Patient Experience and Bowel Preparation for Transvaginal Surgical Management of Vaginal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alicia Ballard, M.D., University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: X100928005
Record Dates: First submitted 2011-08-03; First posted 2011-09-09 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Value of the Bowel Preparation and Diet Change Versus no Intervention; Preoperative Bowel Regimen
Keywords: Bowel Prep; No bowel prep; Vaginal reconstructive or obliterative surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A will have no bowel preparation and be permitted a regular diet the day prior to surgery until midnight.
  Interventions: Other: No bowel prep
- Group B (Active Comparator): Participants in this group will consume a clear liquid diet and perform 2 Fleets enemas in the late afternoon the day before surgery and nothing after midnight.
  Interventions: Other: Clear liquid diet and 2 Fleet's enemas

INTERVENTIONS:
Other: No bowel prep — Participants in this group will have a regular diet and no bowel prep the day prior surgery up until midnight.
  Arms: Group A
Other: Clear liquid diet and 2 Fleet's enemas — Participants in this group will receive a clear liquid diet and 2 Fleets enemas in the late afternoon prior to surgery.
  Other Names: Fleets Saline Enema
  Arms: Group B

SUMMARY:
Preoperative bowel preparation for surgical management of pelvic floor disorders is performed inconsistently, and includes no prep, the use of dietary changes or bowel altering interventions. Retrospective studies of emergency colonic surgery first demonstrated a low rate of infectious complications without a bowel prep. Recently, data supporting the routine use of mechanical cleansing for elective colorectal surgery has demonstrated the surgical outcomes are similar between patients that undergo a bowel preparation versus those that do not, indicating that the long held dogma of mechanical bowel preparation should be used selectively. Despite routine use, there is a paucity of literature addressing the approach to, and/or need for preoperative bowel management at the time of vaginal reconstructive or obliterative surgery. The majority of the pelvic floor disorder population is older, tending to have more bowel dysfunction (especially symptoms of constipation) than younger women.

The aim of this study is to evaluate preoperative bowel management strategy as it relates to the total care of the vaginal surgery patients' intra-and post-operative bowel function and overall patient experience. Two commonly used pre-operative bowel prep strategies: no preoperative bowel prep versus clear fluids and 2-enema prep. The aim is to assess the value of bowel preparation or diet change in vaginal surgery, both from the physician's and patient's point of view. In this pilot study, subjects are randomized to either a clear liquid diet the day prior to surgery with 2 enemas and nothing by mouth (NPO) after midnight, or NPO after midnight without any dietary changes or enemas.

Our aims are:

*Primary - To assess the surgeons' objective intraoperative evaluation of the effects of bowel preparation (adequate visualization, stooling during case, difficulty with bowel handling) *Secondary - (1)To characterize the patients' experience and acceptance of preoperative bowel management regimen versus no preoperative bowel preparation(2) To characterize the patients' postoperative experience and determine if the preoperative bowel regimen affects time to first bowel movement/first normal stool as well as stool experience as recorded by bowel diary (3)Evaluate the incidence of complications between the two groups (4)Characterize other descriptive qualities of the patients' operative experience(duration of case, length of hospital stay)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19
* Female
* Undergoing transvaginal reconstructive surgical intervention for vaginal prolapse (apical suspension and posterior compartment repair required, other concurrent surgery allowed)

Exclusion Criteria:

* Male
* Pregnant, planning pregnancy, or less than 1 year from delivery
* History of total colectomy or prior ileostomy
* Inflammatory bowel disorder (Crohn's disease and ulcerative colitis) formally diagnosed
* Inability to understand written study material (including non-English speaking)
* Inability to give consent
* Presently diagnosed colorectal cancer
* Undergoing chemotherapy and/or radiation
* Chronic constipation suggestive of colonic inertia defined as fewer that 3 stools per week (Rome III guidelines)
* Severe neurological diseases (such as Multiple Sclerosis)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Surgeon assessment of bowel preparation | Will be evaluated at 1 year
  The primary outcome measure will be measured using the surgeon satisfaction questionnaire which is filled out immediately post-op. The surgeon assessment of the bowel preparation and its potential outcome on the surgical field (adequate visualization, stooling during case, and difficulty with bowel handling) will be measured.

SECONDARY OUTCOMES:
Participant experience and acceptance of preoperative bowel management verses no preoperative bowel preparation | Will be evaluated at 1 year
  Participants will complete a patient assessment/satisfaction questionnaire.
Bowel Diary and Bristol Stool Scale | Will be evaluated at 1 year
  Participants will receive 3 seven day bowel diaries,completing one week prior to surgery, and 2 weeks post-operatively. The Bristol Stool Scale is also included as part of the diary and participants are to record each bowel movement during the 3 week period. The information is returned to the physician at the post-operative visit, which occurs approximately 6 weeks after surgery.
Complications between the two groups | Will be evaluated at 1 year
  Any complications that arise will be assessed as they occur and the incidence of complications, if any between the two groups, including wound infection (as defined by erythema, purulent material that was treated with antibiotics, re-operation, or drainage), surgical site breakdown, bowel injury or other unintended injury of adjacent anatomy will be assessed after all the procedures are completed.
Duration of the Case | Will be evaluated at 1 year
  This relates to the overall operative procedure recorded in total operative time.
Length of hospital stay | Will be evaluated at 1 year
  The length of stays will be assessed to gather the average time of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia C Ballard, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, The Kirklin Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ballard AC, Parker-Autry CY, Markland AD, Varner RE, Huisingh C, Richter HE. Bowel preparation before vaginal prolapse surgery: a randomized controlled trial. Obstet Gynecol. 2014 Feb;123(2 Pt 1):232-238. doi: 10.1097/AOG.0000000000000081. PMID 24402594